CLINICAL TRIAL: NCT02261675
Title: Dexmedetomidine Augments Block of Sympathetic Responses to Skin Incision During Sevoflurane Anesthesia in Children
Brief Title: Reduction in MACbar of Sevoflurane by Dexmedetomidine in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cai Li (Other)
Responsible Party: Sponsor-Investigator, Cai Li, Department of Anesthesiology, First Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Macbar DEX
Record Dates: First submitted 2014-10-02; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Children
Keywords: dexmedetomidine; sevoflurane; MAC bar; drug interaction; anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (No Intervention): children undergoing selective lower abdominal surgery received saline before induction
- D1 group (Experimental): children undergoing selective lower abdominal surgery received a bolus dose of 0.5 µg/kg dexmedetomidine followed by a continuous infusion of 0.5 µg/kg /h before induction
  Interventions: Drug: dexmedetomidine
- D2 group (Experimental): children undergoing selective lower abdominal surgery received a bolus dose of 1.0µg/kg dexmedetomidine followed by a continuous infusion of 1.0 µg/kg /h before induction
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — children received intravenous infusion with a bolus dose dexmedetomidine and followed by a continuous infusion before induction. use sevoflurane for induction and a steady-state end-tidal sevoflurane concentration was maintained for at least 15 min before skin incision.
  Other Names: precedex
  Arms: D1 group; D2 group

SUMMARY:
The study was designed to define the interaction of intravenous infusion of dexmedetomidine, an a2-adrenergic agonist, and sevoflurane in children having surgery by using the minimum alveolar concentration which can block adrenergic and cardiovascular responses to incision(MACbar) of sevoflurane as the measure of anesthetic potency.

DETAILED DESCRIPTION:
The investigators observed the effects of different doses of dexmedetomidine on the minimum alveolar concentration of sevoflurane to blockade adrenergic response to surgical incision in 50% of children (MACBAR). And to explore the safety of use of dexmedetomidine in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 2 to 6 yr
* American Society of anesthesiologists I or II
* scheduled to have general anesthesia and to have skin incisions on the abdomen

Exclusion Criteria:

* anemia or abnormal preoperative electrolyte concentrations
* a history of cardiovascular or central nervous system diseases
* a history of pulmonary disease
* known hepatic or renal disease
* a body weight exceeding 50% of the upper limit of ideal body weight for height
* taking drugs with cardiovascular or central nervous system effects
* use of any experimental drug within the past 30 days
* allergy to any drug that may be administered during the study
* exposure to general anesthesia within the previous 7 days
* second- or third-degree atrioventricular block
* taking drugs preoperatively that would interfere with MAC determination(e.g.,opioids or sedatives)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
the end-tidal sevoflurane concentration to blockade adrenergic response to surgical incision in 50% of children (MACBAR) | at once before incision and 5 min period after incision
  A predetermined steady-state end-tidal sevoflurane concentration(4%) was maintained for at least 15 min before skin incision.we observed the change in Mean Blood Pressure or Heart rate to determined the next end-tidal sevoflurane concentration.Followed the modified Dixon up and down method to obtain MACBAR of every child.The MACBAR of sevoflurane and its 95% confidence interval were calculated by Sum Average method.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Ke Liu, Ph.d, Principal Investigator — Departmeng of Anesthesiology, The First Affiliated Hospital, Sun Yat-sen University

REFERENCES:
- [Result] Albertin A, Casati A, Bergonzi P, Fano G, Torri G. Effects of two target-controlled concentrations (1 and 3 ng/ml) of remifentanil on MAC(BAR) of sevoflurane. Anesthesiology. 2004 Feb;100(2):255-9. doi: 10.1097/00000542-200402000-00012. PMID 14739797